CLINICAL TRIAL: NCT03280316
Title: Efficacy Comparison Between Different Management Strategies for Consistent Overactive Bladder (OAB) in Patients With Spinal Vascular Malformations After Surgery
Brief Title: Efficacy Comparison Between Different Management Strategies for Consistent OAB in Patients With SVMs After Surgery
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Principal Investigator, ou tongwen, Director of Urology, Xuanwu Hospital, Beijing
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: otw-20170909
Record Dates: First submitted 2017-09-08; First posted 2017-09-12 (Actual); Last update posted 2020-04-29 (Actual); Status verified 2020-04

CONDITIONS: Spinal Vascular Disorder Nos; Overactive Bladder
Keywords: Spinal Vascular Disorder; Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — Surgical Procedures, Operative; Botulinum Toxins, Type A; Tolterodine Tartrate

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- patients with SVMs undergoing SNM (Experimental): patients with SVMs are of consistent OAB (Overactive Bladder) after surgery and undergo sacral neuromodulation (SNM)
  Interventions: Procedure: surgery; Procedure: sacral neuromodulation
- patients with SVMs receiving BTXA (Experimental): patients with SVMs are of consistent OAB after surgery and accept botulinum toxin A (BTXA) injection
  Interventions: Procedure: surgery; Procedure: botulinum toxin A injection
- patients with SVMs receiving drug (Experimental): patients with SVMs are of consistent OAB (Overactive Bladder) after surgery and accept M receptor antagonist
  Interventions: Procedure: surgery; Drug: M receptor antagonist

INTERVENTIONS:
Procedure: surgery — patients with SVMs receive surgery
Procedure: sacral neuromodulation — sacral neuromodulation (SNM) with InterStimTM
  Arms: patients with SVMs undergoing SNM
Procedure: botulinum toxin A injection — BOTOX
  Arms: patients with SVMs receiving BTXA
Drug: M receptor antagonist — Tolterodine
  Other Names: Tolterodine
  Arms: patients with SVMs receiving drug

SUMMARY:
The investigators' goal is to compare the efficacy of three different management strategies (sacral neuromodulation, botulinum toxin, M receptor antagonist) in treating consistent OAB in patients with SVMs after surgery.

DETAILED DESCRIPTION:
Spinal Vascular malformations (SVMs) are complex neurosurgical lesions and account for 3%-4% of all intradural spinal cord mass lesions, which can influence the function of bladder. The investigators' goal is to compare the efficacy of three different management strategies (sacral neuromodulation, botulinum toxin, M receptor antagonist) in treating consistent OAB (Overactive Bladder) in patients with SVMs after surgery.

ELIGIBILITY:
Inclusion Criteria:

* •Patient diagnosed with spinal vascular diseases including Intradural arteriovenous malformation,Intradural arteriovenous fistula,Dural arteriovenous fistula,Extradural arteriovenous malformation,Paravertebral arteriovenous malformation,Paravertebral arteriovenous fistula,cobbs' syndrome,and other spinal arteriovenous metameric syndromes involve the spinal cord.

  * patient not received surgical or interventional treatment before
  * patient with normal cardiac, renal and hepatic function
  * patient capable of understanding the content of the patient information / Informed Consent Form
  * patient willing and able to participate in the registry
  * patients have consistent OAB after surgery

Exclusion Criteria:

* •patient received surgical treatment or interventional treatment before

  * patient is pregnant
  * patient allergic to iodine
  * patient unable to complete follow-up
  * patient with cerebral lesions
  * patient with other spinal lesions
  * patient with cardiac, renal or hepatic dysfunction

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2023-01 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-12 (Estimated)

PRIMARY OUTCOMES:
bladder function | 3 months and 12 months
  bladder function change in urodynamics

CONTACTS AND LOCATIONS:
Overall Officials: tongwen ou, M.D, Study Director — Xuanwu Hospital, Beijing

IPD SHARING:
Plan to Share IPD: No